CLINICAL TRIAL: NCT04073537
Title: A Randomized, Double-Blind, Multicenter, Phase Ⅲ Study of Anlotinib Hydrochloride Capsule Combined With Chemotherapy Versus Placebo Combined With Chemotherapy in Subjects With Squamous Non-small Cell Lung Cancer
Brief Title: Study of Anlotinib Hydrochloride Capsule Combined With Chemotherapy in Subjects With Squamous Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALTN-03-III-02
Record Dates: First submitted 2019-08-26; First posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Squamous Non-small Cell Lung Cancer
MeSH Terms: interventions — anlotinib; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Anlotinib hydrochloride capsules given orally in fasting conditions , once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21) and paclitaxel 175mg/m2 D1 q3w, carboplatin AUC 5mg/mL/min D1 q3w.
  Interventions: Drug: Anlotinib; Drug: Paclitaxel; Drug: Carboplatin
- Placebo group (Placebo Comparator): Anlotinib hydrochloride placebo given orally in fasting conditions , once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21) and paclitaxel 175mg/m^2 D1 q3w, carboplatin AUC 5mg/mL/min D1 q3w.
  Interventions: Drug: Placebos; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Anlotinib — A multi-target receptor tyrosine kinase inhibitor.
  Arms: Experimental group
Drug: Placebos — Anlotinib blank analog capsule.
  Arms: Placebo group
Drug: Paclitaxel — Paclitaxel 175 mg/m^2 IV on Day 1 of each 21-day cycle.
Drug: Carboplatin — Carboplatin area under the concentration curve (AUC) 5 milligrams per milliliter per minute (mg/mL/min) on Day 1 of each 21-day cycle.

SUMMARY:
Anlotinib hydrochloride is a multi-targeted receptor tyrosine kinase inhibitor that targets angiogenesis-related kinases such as VEGFR1/2/3, FGFR1/2/3, and other tumor-associated kinases involved in cell proliferation such as PDGFRα/β, c-Kit, and Ret have significant inhibitory activities.

ELIGIBILITY:
Inclusion Criteria:

1. Squamous non-small cell lung cancer.
2. A measurable lesion.
3. The disease progression occurs >12 months after the end of the last treatment. 4.18-75 years old ; Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; Life expectancy ≥ 3 months.

5.Adequate laboratory indicators. 6.No pregnant or breastfeeding women, and a negative pregnancy test. 7.Understood and signed an informed consent form.

Exclusion Criteria:

1. The tumor invades the large blood vessels.
2. Central type squamous non-small cell lung cancer.
3. EGFR/ALK gene mutation is positive.
4. Has used EGFR inhibitors and ALK inhibitors.
5. Has other malignant tumors within 5 years.
6. Has a variety of factors affecting oral medications.
7. Symptomatic brain metastasis.
8. Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage.
9. Spinal cord compression.
10. Has received radiotherapy, chemotherapy, surgery less than 4 weeks before randomization.
11. Severe allergies to therapeutic medications.
12. Adverse events caused by previous treatment did not recover to grade 1.
13. Has received major surgical treatment within 4 weeks before randomization.
14. Arteriovenous thrombosis occurred within 6 months.
15. Has drug abuse history that unable to abstain from or mental disorders.
16. Has severe or uncontrolled disease.
17. Participated in other clinical trials within 4 weeks.
18. According to the investigators' judgement.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Estimated)
Dates: Start 2019-10-31 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) evaluated by IRC | up to 24 months
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause; IRC defined as Independent Review Committee.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) evaluated by investigator | up to 24 months
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Overall Survival (OS) | up to 24 months
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.
Overall Response Rate (ORR) | up to 24 months
  Percentage of participants achieving complete response (CR) and partial response (PR).
Disease Control Rate（DCR） | up to 24 months
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of Overall Response (DOR) | up to 24 months
  The time when the patient first achieved complete or partial remission to disease progression.
PFS rate at month 6 | up to 6 months
  The percentage of PFS at month 6.
PFS rate at month 12 | up to 12 months
  The percentage of PFS at month 12.
OS rate at month 6 | up to 6 months
  The percentage of OS at month 6.
OS rate at month 12 | up to 12 months
  The percentage of OS at month 12.
OS rate at month 18 | up to 18 months
  The percentage of OS at month 18.
Adverse Event (AE) | up to 24 months
  Safety data
Serious Adverse Event (SAE) | up to 24 months
  Safety data
Abnormal laboratory test index | up to 24 months
  Safety data

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei